CLINICAL TRIAL: NCT03118804
Title: Weaning From Mechanical Ventilation Guide by Assessment of Lung Tidal Distribution With EIT
Status: Completed | Type: Observational
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, Principal Investigator, Southeast University, China
Other Study IDs: 2016ZDSYLL064-Y01
Record Dates: First submitted 2017-04-09; First posted 2017-04-18 (Actual); Last update posted 2022-11-30 (Actual); Status verified 2022-11

CONDITIONS: Mechanical Ventilation
Keywords: Weaning; Mechanical ventilation; Electrical impedance tomography; Tidal distribution

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Weaning Guide by EIT: Weaning From Mechanical Ventilation Guide by Assessment of Lung Tidal Distribution With EIT
  Interventions: Diagnostic Test: Assessment of Lung Tidal Distribution With EIT

INTERVENTIONS:
Diagnostic Test: Assessment of Lung Tidal Distribution With EIT — Changes of lung tidal distribution during SBT with mechanical ventilation were recorded by EIT can be used to predict weaning success or failure

SUMMARY:
To evaluate whether EELI, RVD, GI were good predictor for weaning from mechanical ventilation

DETAILED DESCRIPTION:
53 patients who ready to wean from mechanical ventilation were included in this study. The changes of lung tidal distribution during SBT with mechanical ventilation by EIT were recorded. Whether EELI, RVD, GI were good predictor for weaning from mechanical ventilation?

ELIGIBILITY:
Inclusion Criteria:

1. Intubated patients age between 18 years old and 80 years old
2. Duration of controlled mechanical ventilation≥ 24 h
3. Patients ready to wean from mechanical ventilation
4. Informed consent

Exclusion Criteria:

1. Pregnant women
2. Patients with malignant tumor
3. High paraplegia, neuromuscular lesions
4. Thoracic deformity, diaphragmatic hernia
5. Patients with ECMO
6. Patient participated in another interventional trial before enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mechanical ventilation admitted to ICU of Zhongda hospital
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-10-18 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Weaning duration | 48 hours
  Time of weaning duration from SBT to weaning from mechanical ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Liu Songqiao, PHD, Principal Investigator — Southeast University
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No